CLINICAL TRIAL: NCT03403621
Title: Double Blind, Single-Center, Randomized, Within Subject Placebo, Phase I Study Evaluating the Effects of Novel Topical Gel in Prevention of Hypertrophic Scar Formation
Brief Title: Hypertrophic Scar Prevention by Novel Topical Gel Application
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding changes.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alexander Meves, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 17-005230
Record Dates: First submitted 2017-12-14; First posted 2018-01-18 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hypertrophic Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Pentamidine

STUDY DESIGN:
Intervention Model Description: All participants will receive two treatments: drug and vehicle. Drug will be applied to one of two treatment sites. Vehicle will be applied to the other site. Treatment sites are distal and proximal end of the incision. Drug will be randomized to treatment site "distal" or "proximal" and masking will be as indicated. A 1-2 cm border zone will remain untreated in the middle of the scar.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will done by the Research Pharmacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topical Pentamidine Isethionate (Experimental): Subjects were randomly assigned to apply topical pentamidine isethionate to either the proximal or distal end of their incision every 48 hours for 4 weeks following surgical scar excision (14-16 treatments).
  Interventions: Drug: Pentamidine Isethionate
- Placebo Control (Placebo Comparator): Subjects were randomly assigned to apply topical placebo to either the proximal or distal end of their incision every 48 hours for 4 weeks following surgical scar excision (14-16 treatments). The subject served as their own control.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentamidine Isethionate — Approximately 1.8 mL single dose delivered as topical formulation containing 2% topical pentamidine in silicone-containing base.
  Other Names: Pentamidine 2% cream
  Arms: Topical Pentamidine Isethionate
Drug: Placebo — No active ingredient. Approximately 1.8 mL single dose delivered as topical silicone compounding base only.
  Other Names: PCCA Pracasil™-Plus (PP)
  Arms: Placebo Control

SUMMARY:
Researchers are trying to find out more about the side effects of topical (applied to the skin) Pentamidine, to determine if it is safe for use in people. They also want to find out if topical use of Pentamidine can help treat hypertrophic scars.

Pentamidine is a medicine that is currently used to treat certain kinds of infection. It is most often given by intravenous (into a vein) or inhalation (through a breathing device). This medication is approved by the U.S. Food and Drug Administration (FDA) for use in these forms.

Everyone in this study will receive topical Pentamidine (TP) in a silicone based gel (PCCA Pracasil Plus). Topical treatment of Pentamidine is still experimental and has not been formally tested for safety or effectiveness in a randomized control trial within the United States. The FDA has allowed the use of topical Pentamidine in this research study.

DETAILED DESCRIPTION:
This study will investigate Pentamidine isethionate, compounded in a silicone-containing base, as adjuvant therapy to surgical scar excision to prevent adverse scarring and enhance skin rejuvenation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertrophic scar by a Mayo Clinic plastic surgeon or dermatologist.
* Target disease or condition: Hypertrophic scar
* Subject with a hypertrophic scar that meet all of the following criteria:

  * Linear scar ≥5 to ≤40 cm in length
  * Present for minimum 6 months
  * Located anywhere in the body except on the face or front of neck
  * Resulting from surgical or traumatic injury, or other scar considered appropriate for surgical excision
* Ability to safely undergo scar excision surgery
* Capacity to provide informed consent
* Ability to comply with protocol
* Subject is judged, by the clinical investigator, to be healthy as evidenced by lack of clinically significant abnormal findings on medical history, physical examination, electrocardiogram, vital signs, and clinical laboratory tests.

Exclusion Criteria:

* Subjects identified as having a keloid or a scar not appropriate for surgical excision
* Subjects who are positive for hepatitis B surface antigen (HbsAg), hepatitis C antibody and HIV as determined in screening the subject's electronic medical record.
* Concurrent use of corticosteroids (including inhaled steroids), cyclooxygenase-2 (COX-2) inhibitors and/or drugs that are strong inhibitors and inducers of cytochrome P450 (CYP) enzymes
* Are immuno-compromised (HIV infected, cancer and other disease affecting the basal immune response)
* Clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurological, psychiatric, immunological, gastrointestinal, hematological, or metabolic disease that is, in the opinion of the investigator, not stabilized or may otherwise impact the results of the study.
* Subjects with renal and hepatic impairment.
* Known allergy or hypersensitivity to the study drug(s) or one of the ingredients of the formulation.
* Any infection or wound in the area to treat including photosensitive dermatosis or inflammatory acne.
* Existence of any surgical, medical or laboratory condition that, in the judgment of the clinical investigator, might interfere with the safety, distribution, metabolism or excretion of the drug
* Participation in another clinical study in the past 30 days or concurrent participation in another clinical trial.
* Patients with poorly controlled diabetes mellitus (HbA1C ≥ 8%), peripheral neuropathy, or known concomitant vascular problems.
* Pregnant or lactating female patients.
* Prisoners.
* Subjects who smoke cigarettes and/or use other tobacco products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Meves, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Scars
Period: Overall Study
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Started | 6; 6 Scars | 6; 6 Scars
Completed | 4; 4 Scars | 4; 4 Scars
Not Completed | 2; 2 Scars | 2; 2 Scars
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants received two treatments: topical pentamidine isethionate and placebo. Participants were randomly assigned to apply topical pentamidine isethionate to either the proximal or distal end of their incision and placebo on the other end of their incision every 48 hours for 4 weeks following surgical scar excision (14-16 treatments).
  Pentamidine Isethionate: Approximately 1.8 mL single dose delivered as topical formulation containing 2% topical pentamidine in silicone-containing base.
  Placebo: No active ingredient. Approximately 1.8 mL single dose delivered as topical silicone compounding base only.
Arm/Group | All Study Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (15.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events
Description: Number of participants to experience serious adverse events as defined as death [due to treatment] or life threatening adverse experience [due to treatment], hospitalization [due to treatment], persistent or significant disability or incapacity [due to treatment], birth defect/anomalies [due to treatment] and tissue necrosis [due to treatment].
Time Frame: 4 weeks post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

2. Secondary Outcome: Adverse Events
Description: Number of participants to experience adverse events as defined as skin infection, skin irritation and wound dehiscence. Skin irritation is scored by local skin reaction (LSR) grading scale. Wound infection is defined by skin that is red, swollen, hot and painful ("calor, dolor, rubor, tumor") [by clinical exam] with or without discharge. Wound dehiscence is defined as a measurable breaking open of the surgical incision along the suture.
Time Frame: 4 weeks post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Number analyzed (Participants) | 6 | 6
Participants | 4 | 5

3. Secondary Outcome: Change in Scar Volume
Description: Ultrasound will be used to quantify hypertrophic scar dimensions (length, width and height) and volume size using cm^3 as the unit of measure.
Time Frame: Baseline (pre-operatively) and at postop week 2 and 4.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Number analyzed (Participants) | 6 | 6
cm^3
  Baseline, 2 weeks post-operative | -0.72 (0.50) | -0.68 (0.52)
  Baseline, 4 weeks post-operative | -0.65 (0.77) | -0.76 (0.52)

4. Secondary Outcome: Change in Scar Fibrosis
Description: Semi-quantitative assessment of scar fibrosis on skin punch biopsy using a scale of none(1) - mild(2) - moderate(3) - severe(4)
Time Frame: Baseline (preoperatively) and 4 weeks post-operatively.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Number analyzed (Participants) | 6 | 6
units on a scale | 1 [1 to 2] | 2 [1 to 2]

5. Secondary Outcome: Change in Scar Sclerosis
Description: Semi-quantitative assessment of scar sclerosis on skin punch biopsy using a scale of none(1) - mild(2) - moderate(3) - severe(4)
Time Frame: Baseline (preoperatively) and 4 weeks post-operatively.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Number analyzed (Participants) | 6 | 6
units on a scale | 0 [0 to 2] | 0 [0 to 0]

6. Secondary Outcome: Change in Scar Angioplasia
Description: Semi-quantitative assessment of scar angioplasia on skin punch biopsy using a scale of none(1) - mild(2) - moderate(3) - severe(4)
Time Frame: Baseline (preoperatively) and 4 weeks post-operatively.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Number analyzed (Participants) | 6 | 6
units on a scale | 0 [-1 to 1] | 0 [-1 to 1]

7. Secondary Outcome: Change in Scar Relative Depth
Description: Semi-quantitative assessment of scar relative depth on skin punch biopsy using a scale of Epidermis(1) - Mid-Reticular Dermis (2) - Deep Dermis(3) - Fat(4)
Time Frame: Baseline (preoperatively) and 4 weeks post-operatively
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Number analyzed (Participants) | 6 | 6
units on a scale | 0 [-1 to 1] | 0 [-1 to 2]

8. Secondary Outcome: Change in Scar Absolute Depth
Description: Measurement of scar absolute depth on skin punch biopsy reporting in millimeters (mm)
Time Frame: Baseline (preoperatively) and 4 weeks post-operatively
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Number analyzed (Participants) | 6 | 6
millimeters | -0.17 (2.26) | 1.34 (2.09)

9. Secondary Outcome: Vancouver Scar Scale (VSS)
Description: The VSS assesses 4 variables: vascularity, height/thickness, pliability, and pigmentation. Scale ranges are as follows. Pigmentation (0=normal, 1=hypopigmentation, 2=hyperpigmentation). Height (0=flat, 1=less than 2 mm, 2=2 to 5 mm, 3=greater than 5 mm). Vascularity (0=normal, 1=pink, 2=red, 3=purple). Pliability (0=normal, 1=supple, 2=yielding, 3=firm, 4=banding,5=contracture). Total score can range from 0 to 13, with 0=normal skin, and 13=severe scarring.
Time Frame: Baseline (preoperatively) and at weeks 2 and 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 5.5 (3.7) | 4.8 (3.6)
  2 weeks | 4.0 (2.2) | 3.5 (3.2)
  4 weeks | 4.8 (2.3) | 5.8 (2.2)
Statistical Analysis 1: Comparison: Topical Pentamidine Isethionate; Baseline versus 2 weeks; Test type: Superiority; p = 0.42, t-test, 2 sided
Statistical Analysis 2: Comparison: Topical Pentamidine Isethionate; Baseline versus 4 weeks; Test type: Superiority; p = 0.72, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo Control; Baseline versus 2 weeks; Test type: Superiority; p = 0.51, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo Control; Baseline versus 4 weeks; Test type: Superiority; p = 0.58, t-test, 2 sided

10. Secondary Outcome: Patient Scar Assessment Scale (PSAS)
Description: The patient scar scale assesses pain, itching, color, stiffness, thickness, and irregularity. The scale rates each variable on a scale from 1 (normal skin) to 10 (worst scar imaginable), with a total possible score ranging from 1 (normal) to 120 (worst scar imaginable).
Time Frame: Baseline (preoperatively) and at weeks 2 and 4.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 39 (8.3) | 43.2 (9.1)
  2 weeks | 27.7 (6.6) | 28.7 (8.9)
  4 weeks | 25.5 (14.8) | 27.0 (11.9)
Statistical Analysis 1: Comparison: Topical Pentamidine Isethionate; Baseline versus 2 weeks; Test type: Superiority; p = 0.03, t-test, 2 sided
Statistical Analysis 2: Comparison: Topical Pentamidine Isethionate; Baseline versus 4 weeks; Test type: Superiority; p = 0.08, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo Control; Baseline versus 2 weeks; Test type: Superiority; p = 0.02, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo Control; Baseline versus 4 weeks; Test type: Superiority; p = 0.007, t-test, 2 sided

11. Secondary Outcome: Observer Scar Assessment Scale (OSAS)
Description: The observer scar assessment scale assesses vascularity, pigmentation, thickness, relief, pliability, and surface area. The scale rates each variable on a scale from 1 (normal skin) to 10 (worst scar imaginable), with a total possible score ranging from 1 (normal) to 120 (worst scar imaginable).
Time Frame: Baseline (preoperatively), 2 weeks, and 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 32.3 (12.8) | 31.2 (13.7)
  2 weeks | 23.5 (10.1) | 23.3 (13.0)
  4 weeks | 23.2 (8.6) | 26.3 (9.9)
Statistical Analysis 1: Comparison: Topical Pentamidine Isethionate; Baseline versus 2 weeks; Test type: Superiority; p = 0.21, t-test, 2 sided
Statistical Analysis 2: Comparison: Topical Pentamidine Isethionate; Baseline versus 4 weeks; Test type: Superiority; p = 0.18, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo Control; Baseline versus 2 weeks; Test type: Superiority; p = 0.33, t-test, 2 sided
Statistical Analysis 4: Comparison: Placebo Control; Baseline versus 4 weeks; Test type: Superiority; p = 0.5, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 3 months on all participants.
Arm/Group | Topical Pentamidine Isethionate | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topical Pentamidine Isethionate (N=6) | Placebo Control (N=6)
Skin Itching (Skin and subcutaneous tissue disorders) | 2 | 4
Skin flaking (Skin and subcutaneous tissue disorders) | 2 | 2
Pustules (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Localized pain (General disorders) | 0 | 1
Bruising (General disorders) | 1 | 0
Wound dehiscence (Surgical and medical procedures) | 1 | 0

LIMITATIONS AND CAVEATS:
Terminated study due to funding changes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT03403621/Prot_SAP_000.pdf